CLINICAL TRIAL: NCT00455091
Title: A Randomization Trial of Adjuvant Lamivudine/ Adefovir Dipivoxil Against Recurrence in Post-operative HBV-related Hepatocellular Carcinoma
Brief Title: A Phase III Study in Post-operative HBV-related Hepatocellular Carcinoma
Status: Terminated | Type: Observational
Why Stopped: No cases enrollment
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Chang Gung Memorial Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Mackay Memorial Hospital (Other); Taichung Veterans General Hospital (Other); Changhua Christian Hospital (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Veterans General Hospital. (Other); Kaohsiung Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: T1206
Record Dates: First submitted 2007-04-02; First posted 2007-04-03 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2009-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Post-operative Hepatocellular Carcinoma.
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — adefovir dipivoxil; Lamivudine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — HBVDNA
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Adefovir Dipivoxil and Lamivudine — Adefovir Dipivoxil 10mg/day x 36 months,Lamivudine 100 mg/day x 18 months#, when HBV DNA =/> 105 copies/mL and ALT > 2.0 x UNL
  Other Names: Hepsera,Zeffix

SUMMARY:
Research Objective and Study End Points To evaluate the anti-HBV as well as HCC recurrence reducing effects of standard (18 months) lamivudine treatment at time of HBV reactivation with hepatitis flare up (HBV DNA > 105 copies/mL and ALT level > 2.0 x UNL) or prophylactic, prolong (36 months) adefovir dipivoxil therapy in post-operative HBsAg(+),< 5 cm HCC patients, and to compare the results of who group with historical controls (T1297, HBsAg+,< 5 cm HCC cohort),in terms of the following endpoints.

1. Primary endpoint:

   the 3-years recurrence rate (excluding those recur within first year).
2. Secondary endpoints:

the first 2 year tumor recurrence rates the recurrence-free survival the overall survival. anti-viral efficacy, i.e. biochemical response and viral response rate. to correlate the changes of viral titer with the clinical outcome in post- operative HCC patients with adjuvant lamivudine or adefovir therapy.

DETAILED DESCRIPTION:
Treatment plan and Randomization scheme:

HBsAg+, HCC< 5 cm with curative resection Stratified with HBV DNA < 105 OR ≥ 105 copies/mL Genotype B or C RANDOMIZATION Prophylactic group Therapeutic control group Adefovir Dipivoxil 10mg/day x 36 months Lamivudine 100 mg/day x 18 months#, when HBV DNA =/> 105 copies/mL and ALT > 2.0 x UNL

* When YMDD mutant present, switch to Adefovir dipivoxil 10mg/day x 24 months. Selection of patients

  1. Eligibility Criteria (1)Histologically proven hepatocellular carcinoma. (2)HCC underwent curative resection within 6 weeks before registration. (3)Grossly, the resection margin should be > 1 cm. (4)Tumors, either single, < 5 cm in size or no more than 3 for size < 3 cm. (5)Patients must have a performance status of ECOG score < 2. (6)Patients must have adequate liver reservation and adequate hemogram. (i)Pugh-Child's Score < 7. (ii)The serum total bilirubin level are < 2 mg/dl. (iii)The prothrombin times are < 3 sec above normal control. (iv)The platelet are > 7.5 x 104 / mm3. (v)The WBC are > 3,000 / mm3. (7)Patient must have serum creatinine < 1.5 mg/dl (8)Cardiac function with NYHA classification < Grade II (9)HBsAg (+) . (10)Signed informed consent.
  2. Ineligibility Criteria

  <!-- -->

  1. Patients who have non-curative resection are not eligible.
  2. Resected HCCs with histologically positive margins are not eligible.
  3. HCCs with radiological evidence of portal vein thrombus are not eligible.
  4. Patients with other systemic diseases which required concurrent usage of glucoticosteroid or immunosuppressant agent(s) are not eligible.
  5. Patients with advanced second primary malignancy are not eligible.
  6. Patients with pregnancy or breast-feeding are not eligible.
  7. Patients with severe cardiopulmonary diseases are not eligible.
  8. Patients with clinically significant psychiatric disorder are not eligible.
  9. Patients who had antineoplastic chemotherapeutic or immuno-therapeutic drugs or corticosteroids within 6 weeks of commencing the protocol are not eligible.
  10. Patients who had prior lamividine and/or adefovir dipivoxil therapy are not eligible.
  11. Anti-HCV positive patients are not eligible. Statistical Consideration

      Sample size:

      With a phase III superior study design, to give an 80% power with a two-sided 5% significance level, 139 patients per each treatment arm should be included in the study. If a 10% drop-out rate is included, totally, 309 patients (155 per study arm) will be required.

      Analysis

      The objectives are as follows:

  1.Primary endpoint: the 3-year recurrence rate (excluding those recur within 1st year)
  1. Second endpoints the recurrence-free survival.
  2. Second endpoints: the overall survival.
  3. Second endpoints: anti-viral efficacy, in terms of sustained biochemical response rate and viral response rate. To correlate the changes of viral titer with the clinical outcome 2 RFS and OS are computed from the date of randomization.

  (1) In analysis of RFS, patients died without disease recurrence will be censored for recurrence at the date of death (2) In analysis of OS, an event is defined as death from any cause. (3) The survival distributions of RFS and OS will be estimated by the Kaplan and Meier method.

  (4) Statistical comparisons of RFS and OS between the two treatment arms will be performed with the log-rank test.

  (5) Cox proportional hazards model will be used to assess the importance of potential prognostic factors, as well as to test the significance of treatment when adjusting for factors [39].

  3.Tumor size, Liver inflammation, viral status, i.e. HBV genotype and DNA titer

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven hepatocellular carcinoma.
2. HCC underwent curative resection within 6 weeks before registration.
3. Grossly, the resection margin should be > 1 cm.
4. Tumors, either single, < 5 cm in size or no more than 3 for size < 3 cm.
5. Patients must have a performance status of ECOG score < 2.
6. Patients must have adequate liver reservation and adequate hemogram.

   * Pugh-Child's Score < 7.
   * The serum total bilirubin level are < 2 mg/dl.
   * The prothrombin times are < 3 sec above normal control.
   * The platelet are > 7.5 x 104 / mm3.
   * The WBC are > 3,000 / mm3.
7. Patient must have serum creatinine < 1.5 mg/dl
8. Cardiac function with NYHA classification < Grade II
9. HBsAg (+) .
10. Signed informed consent.

Exclusion Criteria:

1. Patients who have non-curative resection are not eligible.
2. Resected HCCs with histologically positive margins are not eligible.
3. HCCs with radiological evidence of portal vein thrombus are not eligible.
4. Patients with other systemic diseases which required concurrent usage of glucoticosteroid or immunosuppressant agent(s) are not eligible.
5. Patients with advanced second primary malignancy are not eligible.
6. Patients with pregnancy or breast-feeding are not eligible.
7. Patients with severe cardiopulmonary diseases are not eligible.
8. Patients with clinically significant psychiatric disorder are not eligible.
9. Patients who had antineoplastic chemotherapeutic or immuno-therapeutic drugs or corticosteroids within 6 weeks of commencing the protocol are not eligible.
10. Patients who had prior lamividine and/or adefovir dipivoxil therapy are not eligible.
11. Anti-HCV positive patients are not eligible.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-operative HBV-related Hepatocellular Carcinoma
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2007-05; Primary Completion 2012-04 (Actual); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint: Primary endpoint: the 3-years recurrence rate (excluding those recur within first year). | 6 years

SECONDARY OUTCOMES:
Secondary endpoints: the first 2 year tumor recurrence rates,the recurrence-free survival,the overall survival.anti-viral efficacy. | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, Ph.D., Principal Investigator — National Health Research Institutes, Taiwan; Pei-Jer Chen, Ph.D., Principal Investigator — National Taiwan University Hospital; Miin-Fu Chen, M.D., Study Chair — Chang Gung Memorial Hospital
Locations (8):
- Taiwan (8):
  - Chang-Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Veterans General Hospital-Kaohsiung, Kaohsiung City
  - Chang-Gung Memorial Hospital (Lin-Kou), Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Veterans General Hospital-Taipei, Taipei